CLINICAL TRIAL: NCT04027179
Title: Effects of Tongue Bacterial Dysbiosis Related to Periodontal Therapy on Arterial Pressure Control Based on Salivary Nitrite Availability: a Periodontitis Patients Randomized Controlled Clinical Trial
Brief Title: Tongue Dysbiosis Effects on Arterial Pressure of Periodontitis Patients
Acronym: TODY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Taubate (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE17482019.5.0000.5501
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis; Normal Blood Pressure
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FMS chlorhexidine mouthwash (Experimental): Full-mouth scaling and root planning with manual curettes, 20 ml of 0.12% chlorhexidine gluconate mouthwash irrigation of each periodontal pocket of 5mm of more. Patients will rinse with 0.12% chlorhexidine gluconate mouthwash (20mL/60 seconds/ 2 times a day/ 3 weeks).
  Interventions: Drug: 0.12% chlorhexidine digluconate mouthwash; Procedure: Periodontal instrumentation
- FMS placebo mouthwash (Placebo Comparator): Full-mouth scaling and root planning with manual curettes, 20 ml of placebo mouthwash irrigation of each periodontal pocket of 5mm of more. Patients will rinse with placebo mouthwash (20mL/60 seconds/ 2 times a day/ 3 weeks).
  Interventions: Procedure: Periodontal instrumentation; Drug: Placebo mouthwash
- FMS no mouthwash (Active Comparator): Full-mouth scaling and root planning with manual curettes.
  Interventions: Procedure: Periodontal instrumentation

INTERVENTIONS:
Drug: 0.12% chlorhexidine digluconate mouthwash — 0.12% chlorhexidine digluconate mouthwash (20mL/60 seconds/ 2 times a day/ 3 weeks).
  Arms: FMS chlorhexidine mouthwash
Procedure: Periodontal instrumentation — Full-mouth scaling and root planing with manual curettes within 24 hours in two sections 1 hour each.
Drug: Placebo mouthwash — placebo mouthwash (20mL/60 seconds/ 2 times a day/ 3 weeks).
  Arms: FMS placebo mouthwash

SUMMARY:
Blood pressure control is crucial for individuals' wellbeing. However, many daily aspects such as diet could impair blood pressure control. In addition, many people living under different conditions in different countries are affected by some kind of gum disease. These people experience gingival bleeding, bad breath, teeth mobility and pain. Throughout gum disease development the number of oral germs in the mouth increases including their levels in tongue surface. Oral bacterial are able to convert nitrate widely found in food in nitrite which influences blood pressure. Frequently treatment of gum diseases general combines manual instrumentation with mouthwashes. However, it has been suggested that reduction of oral bacteria by mouthwashes, especially chlorhexidine, is accompanied by decreased conversion of nitrate to nitrite and that this minor nitrite availability would increase blood pressure. Therefore, this is a point to be clarified for patients, physicians and dentists.

This study will investigate the relation between treatment with mouthwashes and blood pressure of patients with destructive gum disease based on nitrite levels in saliva, bacterial levels in tongue and values of arterial blood pressure which will be monitored over 6 months. In addition, usual clinical parameters and alteration of oral cells' DNA will be also monitored overtime. Patients will be treated under local anesthesia and manual instrumentation within 24 hours. They will receive oral care products too. There will be 3 treatment groups (manual instrumentation + chlorhexidine mouthwash [2 times a day for 3 weeks], manual instrumentation + placebo mouthwash [2 times a day for 3 weeks] and manual instrumentation + no mouthwash) and 2 dental appointments before treatment. After treatment, patients will be examined at 7, 14, 21, 90 and 180 days. Saliva, plaque and cell sampling will be fast and by no invasive methods.

ELIGIBILITY:
Inclusion Criteria:

* 12 natural teeth; chronic periodontitis stages II and III; no systemic medication; non smokers; normal blood pressure; no mouthwash regular use; antibiotics > 3 months prior to study; dental treatment > 3 months prior to study.

Exclusion Criteria:

- known alergy to chlorhexidine; removable prosthodontics apparatus; pregnant and breast feeding women.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy - comparative tongue bacterial counts | Baseline and 3 months
  Changes of Veillonella, Streptococcus, Neisseria, Fusobacterium and Acytinomyces counts in samples from tongue dorsal

SECONDARY OUTCOMES:
Safety - comparative nitrite levels in saliva | Baseline and 3 months
  Differences in mean nitrite levels from saliva samples pre- and post-treatment
Safety - Percentage of hypertension episodes | Baseline and 3 months
  Changes in the percentage of hypertension episode
Safety - status of DNA methylation in oral cells | Baseline and 3 months
  Mean changes of DNA methylation statuses in oral cells
Efficacy - Percentage of periodontal pockets | Baseline and 6 months
  Changes in the percentage of deep periodontal pockets

CONTACTS AND LOCATIONS:
Locations (1):
- University of Taubate - Nucleus of periodontal research, Taubaté, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No